CLINICAL TRIAL: NCT02927093
Title: Neonatal, Clinical and Neurodevelopmental Outcome of Neonates Hospitalized for Neonatal Hyperbilirubinemia Reaching Exchange Transfusion Threshold in a Remote Setting Along the Thai-Myanmar Border
Brief Title: Clinical and Developmental Outcomes of Babies Who Became Yellow in the First Month of Life
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU 1605
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: neonates with NH reaching exchange transfusion threshold
- Control: neonates with NH within moderate threshold of the phototherapy charts

SUMMARY:
The Shoklo Malaria Research Unit (SMRU) provides care to refugees and migrant populations along the Thai-Burma border since 1986. Services include antenatal and birthing care, with 2,500 births per year and Special Care Baby Units (SCBU) set up in 2008; all medical records including clinical and laboratory data are archived. The treatment of neonatal jaundice is based on treatment thresholds adapted from the neonatal jaundice guidelines, published by the Royal College of Obstetricians and Gynaecologists, UK. Total serum bilirubin (SBR) is done at regular intervals to monitor neonatal hyperbilirubinemia (NH) evolution, following SMRU guidelines. The SCBU have been set up to provide intensive care for neonates in a resource constrained setting and don't have equipment for assisted ventilation other than oxygen therapy. Neonates presenting with high serum bilirubin levels and/or clinical signs of acute bilirubin encephalopathy (ABE) cannot receive exchange transfusion on site and have to be referred to the Thai general hospital one hour drive from the clinics; and, for those neonates surviving, there has not been a systematic follow-up of their growth and neurodevelopment.

The study will consist of a matched case-control series and a retrospective review of SCBU charts of neonates with NH reaching exchange transfusion threshold. The SCBU database will be searched for neonates born at ≥ 28 weeks of gestation hospitalized for phototherapy between January 2009 and December 2014; charts will be manually researched to identify study participants which will be classified as NH reaching exchange transfusion threshold (cases) or as NH within moderate threshold (controls). Additionally neurological signs compatible with ABE will be searched in the clinical notes and coded as present/absent. Cases discharged alive from the SCBU will be traced back to evaluate their clinical and neurocognitive long term outcome. Each case will be matched with a moderate NH control from the same clinic, sex, gestational age and season of birth and hospitalized within the same month.

The results of this study will help to improving the clinical care during the neonatal period and to developing a guideline for a better follow-up of children with NH reaching exchange transfusion threshold.

DETAILED DESCRIPTION:
The study will consist of a matched case-control series and a retrospective review of SCBU charts of neonates with NH reaching exchange transfusion threshold.

The SCBU database will be searched for neonates born at ≥ 28 weeks of gestation hospitalized for phototherapy between January 2009 and December 2014. The SCBU charts of these neonates will be manually researched to identify study participants which will be classified as NH reaching exchange transfusion threshold (cases) or as NH within moderate threshold (controls). Additionally neurological signs compatible with ABE that would likely be reported by the clinical staff will be searched in the clinical notes and coded as present/absent; those signs are: sleepiness, irritability, apnea, convulsions, abnormal position/tone, and abnormal cry. Those charts will be included into the cases.

Cases discharged alive from the SCBU will be traced back to evaluate their clinical and neurocognitive long term outcome. Each case will be matched with a moderate NH control from the same clinic, sex, gestational age and season of birth and hospitalized within the same month.

Both will be examined clinically and findings reported on a standardized forms, their visual function will be tested using the Cardiff acuity and contrast cards and their neurocognitive development will be assessed using the Griffiths Mental Development Scales-Extended revised.

Maternal demographics and additional birth variables (i.e. birth asphyxia, type of delivery, breastfeeding) will be extracted from the antenatal care database and added to the selected cases; laboratory results (G6PD deficiency, ABO incompatibility, haematocrit) are stored in the SCBU database and will be retrieved. The general characteristics, the trajectory of SBR, and the neonatal outcome will be described.

ELIGIBILITY:
Inclusion Criteria:

Cases

Liveborn, singleton, ≥28 weeks gestation, hospitalized at SMRU SCBU presenting one or more of the following criteria:

* Two consecutive SBR measures above the exchange transfusion threshold of the phototherapy charts for gestational age
* SBR levels rising > 8.5 µmol/L per hour
* One or more neurological signs compatible with ABE in the absence of other known neurological condition and in the presence of confirmed NH

Controls

Liveborn singleton, ≥28 weeks gestation, hospitalized at SMRU SCBU presenting all of the following criteria:

* At least one SBR between the moderate and the severe threshold of the phototherapy charts for gestational age
* No SBR above the severe threshold at any time point
* No reported abnormal neurological signs (i.e. convulsions, abnormal cry or tone)

Each case who has been discharged alive from the SCBU will be matched to one control from the same clinic, sex, gestational age, season of birth and hospitalized within the same month and the clinical and neurodevelopment of both children will be conducted once.

Exclusion Criteria:

* Stillborn
* Twins
* Liveborn < 28 weeks gestation
* Major congenital malformation
* Liveborn singleton, ≥28 weeks gestation, hospitalized outside SMRU SCBU
* Liveborn singleton, ≥28 weeks gestation, hospitalized at SMRU SCBU without SBR done or with all SBR below the moderate threshold of the phototherapy charts for gestational age

Min Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Liveborn, singleton, ≥28 weeks gestation, hospitalized at SMRU SCBU, from 1st January 2009 to 31st December 2014 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Visual Function Scores | 8 years
  The odds ratio of visual function scores between survivors of NH reaching exchange transfusion threshold and those with moderate NH
Neurodevelopmental scores | 8 years
  The odds ratio of neurodevelopmental scores between survivors of NH reaching exchange transfusion threshold and those with moderate NH
Clinical status | 8 years
  The clinical status between survivors of NH reaching exchange transfusion threshold and those with moderate NH

SECONDARY OUTCOMES:
Mortality rate | 8 years
  The mortality rate among neonates with NH reaching exchange transfusion threshold
Proportion of neonates with ABE | 8 years
  The proportion of neonates with ABE among those with NH reaching exchange transfusion threshold
Proportion of neonates with G6PD deficiency | 8 years
  The proportion of neonates with G6PD deficiency present among neonates with NH reaching exchange transfusion threshold
Proportion of neonates with ABO incompatibility | 8 years
  The proportion of neonates with ABO incompatibility present among neonates with NH reaching exchange transfusion threshold
Proportion of neonates with polycythaemia | 8 years
  The proportion of neonates with polycythaemia present among neonates with NH reaching exchange transfusion threshold
Proportion of neonates with birth trauma | 8 years
  The proportion of neonates with birth trauma present among neonates with NH reaching exchange transfusion threshold
Proportion of neonatal sepsis | 8 years
  The proportion of neonatal sepsis present among neonates with NH reaching exchange transfusion threshold
Proportion of neonates with prematurity | 8 years
  Proportion of neonates with prematurity present among neonates with NH reaching exchange transfusion threshold

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in the database and may be shared with other researchers in the future, however, data will be anonymous and the researchers will not know the participant identity.